CLINICAL TRIAL: NCT00867035
Title: Bad Breath Response to Tongue Scraper and Rinses, a Double-blind, Randomized, Parallel Group Clinical Trial.
Brief Title: Bad Breath Response to Tongue Scraper and Rinses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PGP1
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Results first posted 2013-05-16 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Halitosis
MeSH Terms: conditions — Halitosis | interventions — chlorine dioxide; chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chlorhexidine gluconate and scraper (Active Comparator): The intervention was accomplished by subject after instructions from investigator: twice a day a tongue scraper was used with 4 or more strokes, followed by 20ml of 0.12% chlorhexidine gluconate mouthwash used for 30 sec, for one week.
  Interventions: Drug: Chlorhexidine gluconate and scraper
- Chlorine dioxide and scraper (Experimental): The intervention was accomplished by subject after instructions by investigator: twice a day the scraper was used for 4 strokes then 20ml 0.1% stabilized chlor8ine dioxide rinse for 30sec, for one week.
  Interventions: Drug: Chlorine dioxide and scraper

INTERVENTIONS:
Drug: Chlorine dioxide and scraper — 20ml of mouthwash used for 30sec as adjunct to tongue scraper twice a day
  Other Names: "CloSYS"
  Arms: Chlorine dioxide and scraper
Drug: Chlorhexidine gluconate and scraper — The intervention was accomplished by subject after instructions by investigator: twice a day the scraper was used for 4 strokes then 20ml 0.12% chlorhexidine gluconate rinse for 30sec, for one week.
  Other Names: "Peridex"
  Arms: Chlorhexidine gluconate and scraper

SUMMARY:
Medical center personnel were screened organoleptically for bad breath by 2 investigators using Rosenberg scale 0-5, and measurement of breath sample in portable gas chromatograph. With a threshold score of 2 or more, or 75parts per billion(ppb) hydrogen sulfide(H2S), subjects invited to enter clinical trial of the mechanical effect of daily tongue scraping with the adjunctive use of 0.12% chlorhexidine gluconate mouthwash or 0.1% stabilized chlorine dioxide mouthwash. Subjects randomly assigned in double-blind trial for one week. The null hypothesis is there will be no difference between the two rinses as adjuncts to tongue scraping.

DETAILED DESCRIPTION:
Subjects in trial had oral and periodontal exam and scored the Ramfjord teeth(#3, 9, 12, 19, 25, 28) for Plaque Index(PlI), Gingival Index(GI), probing depth (PD), recession. A tongue coating index is scored and sample of coating on dorsum taken for culture of total viable count and percentage of black sulfide-producing colonies on anaerobe agar with lead acetate added. Subjects given hygiene instruction and instruction on use of scraper, then rinse with 20ml assigned mouthwash 30sec. Breath assessed by organoleptic means and mouth air sample concentration of hydrogen sulfide, methyl mercaptan in portable gas chromatograph at 0, 1, 2, and 4 hours. Subjects use scraper and mouthwash twice daily for one week and return for final exam.

ELIGIBILITY:
Inclusion Criteria:

* Adult with threshold score of 2 on organoleptic halitosis evaluation

Exclusion Criteria:

* Taking another experimental drug, or antibiotic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milton R Wirthlin, DDS, Principal Investigator — University of California, San Francisco
Locations (1):
- UCaliforniaSF, San Francisco, California, United States

REFERENCES:
- [Result] Wirthlin MR, Im T, Ellis RR, Hoover CI. Effect of tongue scraper and rinses on bad breath, a double-blind, randomized, parallel group clinical trial. J West Soc Periodontol Periodontal Abstr. 2011;59(3):67-73. No abstract available. PMID 22141237

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening in dental clinic March 2008-March 2009. With organoleptic(OLT)score of 2 or more, or 75parts per billion(ppb) hydrogen sulfide(H2S), subjects invited to enter clinical trial. Subjects numbered in sequence from a computer-generated table of random numbers.
Pre-assignment Details: Exclusions: 1)Inability to return for evaluation, 2)inability to follow directions, 3) afflicted with systemic disease involving volatile sulfur compounds (VSC), 4)currently taking antibiotics, 5) using medicine in syrup form, 6) advanced periodontal disease, 7) smoker.
Groups:
- Chlorine Dioxide Rinse and Tongue Scraper: 20ml of a stabilized 0.1% chlorine dioxide mouthrinse is used after use of tongue scraper twice a day
- Chlorhexidene Rinse and Tongue Scraper: 20ml of 0.12% chlorhexidine gluconate mouthrinse is used after tongue scraping twice a day
Period: Baseline to 1 Hour
Arm/Group | Chlorine Dioxide Rinse and Tongue Scraper | Chlorhexidene Rinse and Tongue Scraper
Started | 13 | 9
Completed | 12 | 8
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Baseline to 2 Hours
Arm/Group | Chlorine Dioxide Rinse and Tongue Scraper | Chlorhexidene Rinse and Tongue Scraper
Started | 12 | 8
Completed | 12 | 8
Not Completed | 0 | 0
Period: Baseline to 4 Hours
Arm/Group | Chlorine Dioxide Rinse and Tongue Scraper | Chlorhexidene Rinse and Tongue Scraper
Started | 12 | 8
Completed | 12 | 8
Not Completed | 0 | 0
Period: Baseline to 1 Week
Arm/Group | Chlorine Dioxide Rinse and Tongue Scraper | Chlorhexidene Rinse and Tongue Scraper
Started | 12 | 8
Completed | 11 | 8
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chlorine Dioxide Rinse and Tongue Scraper | Chlorhexidene Rinse and Tongue Scraper | Total
Number analyzed (Participants) | 13 | 9 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 9 | 22
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 9 | 6 | 15
Region of Enrollment [Number; unit: participants]
  United States | 13 | 9 | 22
Rosenberg score of 2 or more [Number; unit: participants] — The Rosenberg scale is validated and is scored 0-5 with 0= no bad breath, 5=worst bad breath. A score of 2 is the threshold at which bad breath is determined
  participants | 13 | 9 | 22

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Rosenberg Score at Indicated Time Points
Description: 2 investigators are trained to evaluate smell using the Rosenberg scale which measures foul smelling breath. The Rosenberg scale is validated and is scored 0-5 with 0= no bad breath, 5=worst bad breath. A score of 2 is the threshold at which bad breath is determined.
Time Frame: baseline, 1 hour, 2 hours, 4 hours, 1 week
Population: two judges score breath odor by Rosenberg scale 0 to 5. Score of 2 is threshold for malodor. participants randomly assigned, ITT.
Measure: Number; unit: percentage of participants
Arm/Group | Chlorine Dioxide Rinse and Tongue Scraper | Chlorhexidene Rinse and Tongue Scraper
Number analyzed (Participants) | 13 | 9
percentage of participants
  Percentage with score of 2 or 3 at Baseline | 96 | 74
  Percentage with score of 0 or 1 at 1 hour | 79 | 100
  Percentage with score of 0 or 1 at 2 hours | 79 | 94
  Percentage with score of 0 or 1 at 4 hours | 54 | 81
  Percentage with score of 0 or 1 at 1 week | 64 | 81
Statistical Analysis 1: Comparison: Chlorine Dioxide Rinse and Tongue Scraper; Rosenberg scores compared baseline to 1 hour by Mann-Whitney U test; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Chlorhexidene Rinse and Tongue Scraper; mann whitney u to compare rosenberg score baseline to 1 hour; Test type: Superiority or Other; p < .001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Chlorine Dioxide Rinse and Tongue Scraper; baseline to 2 hours; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Chlorine Dioxide Rinse and Tongue Scraper; baseline to 4 hours; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Chlorine Dioxide Rinse and Tongue Scraper; baseline to 1 week; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Chlorhexidene Rinse and Tongue Scraper; baseline to 2 hours; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Chlorhexidene Rinse and Tongue Scraper; baseline to 4 hours; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Chlorhexidene Rinse and Tongue Scraper; baseline to 1 week; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Concentration of Hydrogen Sulfide (H2S) in Mouth Air at 1 Hour
Description: Using portable gas chromatograph
Time Frame: 1hr
Population: ITT
Measure: Mean (Standard Deviation); unit: parts per billion (ppb)
Arm/Group | Chlorine Dioxide Rinse and Tongue Scraper | Chlorhexidene Rinse and Tongue Scraper
Number analyzed (Participants) | 13 | 9
parts per billion (ppb) | 10.1 (18.6) | 9.12 (13.9)
Statistical Analysis 1: Comparison: Chlorine Dioxide Rinse and Tongue Scraper vs Chlorhexidene Rinse and Tongue Scraper; Concentrations of H2S in mouth air at 1 hour analyzed between groups; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

3. Secondary Outcome: Concentration of Hydrogen Sulfide (H2S) in Mouth Air at 2 Hours
Description: Using portable gas chromatograph
Time Frame: 2hr
Population: ITT
Measure: Mean (Standard Deviation); unit: parts per billion (ppb)
Arm/Group | Chlorine Dioxide Rinse and Tongue Scraper | Chlorhexidene Rinse and Tongue Scraper
Number analyzed (Participants) | 12 | 8
parts per billion (ppb) | 12.7 (12.9) | 3.88 (7.57)
Statistical Analysis 1: Comparison: Chlorine Dioxide Rinse and Tongue Scraper vs Chlorhexidene Rinse and Tongue Scraper; Concentrations of H2S in mouth air at 2 hours analyzed between groups. Each time point was compared between groups by Students t test; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

4. Secondary Outcome: Concentration of Hydrogen Sulfide (H2S) in Mouth Air at 4 Hours
Description: Using portable gas chromatograph
Time Frame: 4 hours
Population: ITT
Measure: Mean (Standard Deviation); unit: parts per billion (ppb)
Arm/Group | Chlorine Dioxide Rinse and Tongue Scraper | Chlorhexidene Rinse and Tongue Scraper
Number analyzed (Participants) | 12 | 8
parts per billion (ppb) | 12.7 (16.1) | 7.0 (9.99)
Statistical Analysis 1: Comparison: Chlorine Dioxide Rinse and Tongue Scraper vs Chlorhexidene Rinse and Tongue Scraper; Concentrations of H2S in mouth air at 4 hours analyzed between groups; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

5. Secondary Outcome: Concentration of Hydrogen Sulfide (H2S) in Mouth Air at 1 Week
Description: Using portable gas chromatograph
Time Frame: 1 week
Population: ITT
Measure: Mean (Standard Deviation); unit: parts per billion (ppb)
Arm/Group | Chlorine Dioxide Rinse and Tongue Scraper | Chlorhexidene Rinse and Tongue Scraper
Number analyzed (Participants) | 11 | 8
parts per billion (ppb) | 9.17 (13.1) | 20.2 (29.6)
Statistical Analysis 1: Comparison: Chlorine Dioxide Rinse and Tongue Scraper vs Chlorhexidene Rinse and Tongue Scraper; Concentrations of H2S in mouth air at 1 week analyzed between groups. Each time point was compared between groups by Students t test; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

6. Secondary Outcome: Concentration of Methyl Mercaptan (MM) in Mouth Air at 1 Hour
Description: Using portable gas chromatograph
Time Frame: 1 hour
Population: ITT
Measure: Mean (Standard Deviation); unit: parts per billion (ppb)
Arm/Group | Chlorine Dioxide Rinse and Tongue Scraper | Chlorhexidene Rinse and Tongue Scraper
Number analyzed (Participants) | 13 | 9
parts per billion (ppb) | 17.5 (27.0) | 36.0 (51.0)
Statistical Analysis 1: Comparison: Chlorine Dioxide Rinse and Tongue Scraper vs Chlorhexidene Rinse and Tongue Scraper; Concentrations of MM in mouth air at 1 hour analyzed between groups; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

7. Secondary Outcome: Concentration of Methyl Mercaptan (MM) in Mouth Air at 2 Hours
Description: Using portable gas chromatograph
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: parts per billion
Arm/Group | Chlorine Dioxide Rinse and Tongue Scraper | Chlorhexidene Rinse and Tongue Scraper
Number analyzed (Participants) | 12 | 8
parts per billion | 14.5 (27.4) | 23.9 (33.5)
Statistical Analysis 1: Comparison: Chlorine Dioxide Rinse and Tongue Scraper vs Chlorhexidene Rinse and Tongue Scraper; Concentrations of MM in mouth air at 2 hours analyzed between groups. Each time point was compared between groups by Students t test; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

8. Secondary Outcome: Concentration of Methyl Mercaptan (MM) in Mouth Air at 4 Hours
Description: Using portable gas chromatograph
Time Frame: 4 hours
Population: ITT
Measure: Mean (Standard Deviation); unit: parts per billion
Arm/Group | Chlorine Dioxide Rinse and Tongue Scraper | Chlorhexidene Rinse and Tongue Scraper
Number analyzed (Participants) | 12 | 8
parts per billion | 14.4 (21.2) | 6.88 (9.42)
Statistical Analysis 1: Comparison: Chlorine Dioxide Rinse and Tongue Scraper vs Chlorhexidene Rinse and Tongue Scraper; Concentrations of MM in mouth air at 4 hours analyzed between groups. Each time point was compared between groups by Students t test; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

9. Secondary Outcome: Concentration of Methyl Mercaptan (MM) in Mouth Air at 1 Week
Description: Using portable gas chromatograph
Time Frame: 1 week
Population: ITT
Measure: Mean (Standard Deviation); unit: parts per billion
Arm/Group | Chlorine Dioxide Rinse and Tongue Scraper | Chlorhexidene Rinse and Tongue Scraper
Number analyzed (Participants) | 11 | 8
parts per billion | 9.75 (16.6) | 2.12 (3.64)
Statistical Analysis 1: Comparison: Chlorine Dioxide Rinse and Tongue Scraper vs Chlorhexidene Rinse and Tongue Scraper; Concentrtations of MM in mouth air at 1 week analyzed between groups. Each time point was compared between groups by Students t test; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

10. Secondary Outcome: Number of Bacteria on Tongue at 1 Week
Description: Total viable count(TVC) in colony forming units(CFU) on anaerobe agar
Time Frame: 1 week
Population: ITT
Measure: Mean (Standard Deviation); unit: colony forming units (CFU)
Arm/Group | Chlorine Dioxide Rinse and Tongue Scraper | Chlorhexidene Rinse and Tongue Scraper
Number analyzed (Participants) | 11 | 8
colony forming units (CFU) | 15500000 (25400000) | 28400000 (65400000)
Statistical Analysis 1: Comparison: Chlorine Dioxide Rinse and Tongue Scraper vs Chlorhexidene Rinse and Tongue Scraper; Counts of colony forming units from swab of 1square centimeter area on tongue at 1 week cultured on anaerobe plates for 1 week analyzed between groups; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

11. Secondary Outcome: Percentage of Sulfide-producing Black Colonies Out of Total Viable Count(TVC) on Anaerobe Agar Containing Lead Acetate
Time Frame: 1 week
Population: ITT
Measure: Mean (Standard Deviation); unit: percentage black colonies
Arm/Group | Chlorine Dioxide Rinse and Tongue Scraper | Chlorhexidene Rinse and Tongue Scraper
Number analyzed (Participants) | 11 | 8
percentage black colonies | 43.1 (22.8) | 27.8 (15.6)
Statistical Analysis 1: Comparison: Chlorine Dioxide Rinse and Tongue Scraper vs Chlorhexidene Rinse and Tongue Scraper; Percentage of black colonies out of Total Viable Count cultured on anaerobe agar with lead acetate. Black colonies are those producing sulfides (H2S, MM)and creating black lead sulfide. Analyzed between groups. Groups compared at baseline and 1 week; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Chlorine Dioxide Rinse and Tongue Scraper | Chlorhexidene Rinse and Tongue Scraper
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/9
Other Adverse Events (participants affected / at risk) | 0/13 | 1/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chlorine Dioxide Rinse and Tongue Scraper (N=13) | Chlorhexidene Rinse and Tongue Scraper (N=9)
Effect on taste threshhold (Nervous system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Total number of subjects is less than the desired 50 persons; dimethyl sulfide measures distorted by materials in syringes; accuracy of portable gas chromatograph a concern.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes